CLINICAL TRIAL: NCT02135731
Title: APHID- Sensitivity and Specificity of a Medication Reconciliation Technology - A Primary Care Randomized Controlled Trial
Brief Title: APHID- Primary Care Accuracy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blake Lesselroth (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Blake Lesselroth, Director, Portland Patient Safety Center of Inquiry, Portland VA Medical Center
Organization: Portland VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 08-0308
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Medication Review

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paper (No Intervention): Usual care -medication review on paper
- Computer (Experimental): Medication review software with pictures
  Interventions: Other: Medication review software with pictures

INTERVENTIONS:
Other: Medication review software with pictures — The intervention is a self-service software program that displays each prescription on screen along with an image of the pharmaceutical product. Patients must use response buttons to describe adherence patterns and to advance through the questionnaire items.
  Arms: Computer

SUMMARY:
We are studying patients' abilities to correctly identify the prescription medications they are taking. We are interested in understanding what tools will help patients correctly identify their medications. People participating in this study will be asked to either review a paper printout of their medication list or a computer program with their medications. The program will show the names and pictures of the medications. In either situation, participants will be asked to indicate if they are taking the medications as prescribed. We will then compare reported adherence between each medication review process. Participation may help the program developers improve the product.

DETAILED DESCRIPTION:
The trial compares a paper-based medication adherence questionnaire to an electronic medication adherence questionnaire. Results from each arm will be compared to the ambulatory medication list on file with the clinic and a separate medication review interview conducted by a trained clinician. We intend to compare adherence patterns and medication use discrepancy rates between each approach. This data will help us to determine what strategies work best to solicit an accurate medication history from the patient.

ELIGIBILITY:
Inclusion Criteria:

* Veteran with Primary Care appointment at Portland VA
* Three or more medications in medication profile

Exclusion Criteria:

* Visual impairment
* Upper extremity neuromuscular impairment
* Cognitive impairment
* Unable to speak and read English
* Never been seen at a VA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of medication discrepancies from the reference standard | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Blake Lesselroth, MD, MBI, Principal Investigator — PVAMC
Locations (1):
- Portland VAMC, Portland, Oregon, United States

REFERENCES:
- [Background] Lesselroth BJ, Felder RS, Adams SM, Cauthers PD, Dorr DA, Wong GJ, Douglas DM. Design and implementation of a medication reconciliation kiosk: the Automated Patient History Intake Device (APHID). J Am Med Inform Assoc. 2009 May-Jun;16(3):300-4. doi: 10.1197/jamia.M2642. Epub 2009 Mar 4. PMID 19261949
- [Background] Lesselroth BJ, Adams K, Tallett S, Wood SD, Keeling A, Cheng K, Church VL, Felder R, Tran H. Design of admission medication reconciliation technology: a human factors approach to requirements and prototyping. HERD. 2013 Spring;6(3):30-48. doi: 10.1177/193758671300600304. PMID 23817905
- [Background] Lesselroth BJ, Holahan PJ, Adams K, Sullivan ZZ, Church VL, Woods S, Felder R, Adams S, Dorr DA. Primary care provider perceptions and use of a novel medication reconciliation technology. Inform Prim Care. 2011;19(2):105-18. doi: 10.14236/jhi.v19i2.802. PMID 22417821
- [Derived] Lesselroth BJ, Adams K, Church VL, Tallett S, Russ Y, Wiedrick J, Forsberg C, Dorr DA. Evaluation of Multimedia Medication Reconciliation Software: A Randomized Controlled, Single-Blind Trial to Measure Diagnostic Accuracy for Discrepancy Detection. Appl Clin Inform. 2018 Apr;9(2):285-301. doi: 10.1055/s-0038-1645889. Epub 2018 May 2. PMID 29719884